CLINICAL TRIAL: NCT06644989
Title: Impact of Spencer's Technique of the Hip on Hip Range of Motion in Recreational Runners
Brief Title: Impact of Osteopathic Manipulative Therapy on Hip Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lake Erie College of Osteopathic Medicine (Other)
Collaborators: Lake Erie College of Osteopathic Medicine (LECOM) (Unknown)
Responsible Party: Principal Investigator, Rebecca Steiner, Ph.D., Assistant Professor of Biochemistry and Genetics, Lake Erie College of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Protocol 31-085
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Runners
Keywords: Osteopathic Manipulative Therapy; Spencer Technique
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham Comparator (Sham Comparator): Half of Participants receive Spencer technique and half of participants received a sham treatment.
  Interventions: Other: Sham (No Treatment)
- Experimental (Experimental): Half of Participants receive Spencer technique and half of participants received a sham treatment.
  Interventions: Procedure: Spencer Technique

INTERVENTIONS:
Procedure: Spencer Technique — Spencer technique on the hip
  Arms: Experimental
Other: Sham (No Treatment) — Spencer technique position but no pressure
  Arms: Sham Comparator

SUMMARY:
One way for runners to improve their performance and remain injury free is to preserve and improve joint mobility, especially at the hips. The femoroacetabular joints are a pivotal part of the running gait allowing the athlete to fully extend their leg to generate sufficient force in each stride. Improving hip range of motion can help reduce or prevent groin pain, make the runner more comfortable while running, improve running longevity, and prevent injuries. Thus, it is clear that a runner's commitment to improving the range of motion of their hips is crucial for both the enhancement of their performance and prevention of injury. Researchers assessed how the hip, and its biomechanics, can be impacted by Osteopathic medical treatment.

The primary research question investigated is how Spencer Technique for the hip impacts femoral acetabular active range of motion (AROM) in flexion, extension, abduction, adduction, internal rotation, and external rotation in those training 4 weeks for a 5K race. This study investigated the effect that 4 weeks of twice weekly, bilateral, Spencer Technique treatment had on femoroacetabular range of motion. During this 4-week period participant exercise and stretching habits in preparation for the 5k race were recorded.

ELIGIBILITY:
Inclusion Criteria:

* All LECOM-Bradenton students will be included in recruitment.

Exclusion Criteria:

* Subjects will be excluded from this research study if they cannot sign an informed consent. Additionally, subjects will be excluded if they are:

  * Pregnant or plan to become pregnant
  * Have a past medical history including:

    * Skin disorders or open wounds precluding skin contact
    * Neurological symptoms (i.e. numbness, tingling, weakness)
    * Recent bone fracture
    * Recent lower extremity ligamentous sprain
    * Recent lower extremity muscle strain
    * Adhesive capsulitis of the hip joint
    * Osteoarthritis of the lower extremity
    * Rheumatoid arthritis
    * History of hip or knee arthroplasty
    * 1 year history of any lower extremity surgery
    * Gout
    * Iliotibial band syndrome
    * Legg-Calve-Perthes disease
    * Slipped capital femoral epiphysis
    * Hip dysplasia
    * Avascular necrosis of the hip
    * Chronic hip bursitis
    * Hip dislocation
    * Osteoporosis/osteopenia
    * Severe Femoroacetabular impingement
    * Use of heel lift due to leg length discrepancy
    * Immunosuppressive syndromes
    * Radiation or chemotherapy within the past 3 years
    * Congestive heart failure
    * Unable to complete a 5 kilometer race after the 4 weeks of training
    * Down syndrome
    * Have been told by a physician or other medical professional that you should not participate in aerobic training activities.
    * Have medication changes in the last month
    * Run 30+ miles per week regularly

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Range of Motion | 4 weeks
  Hip range of motion (flexibility) is measured to monitor changes in flexibility

CONTACTS AND LOCATIONS:
Locations (1):
- LECOM, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided